CLINICAL TRIAL: NCT00230711
Title: Physical Activity Promotion In Cancer Follow-up Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: American Cancer Society; RSGP-03-423
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2005-09

CONDITIONS: Breast Cancer
Keywords: Physical activity; Cancer follow-up care
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

ARMS (2):
- Exercise Counseling (Experimental)
  Interventions: Behavioral: Physical activity counseling
- Contact Control (Placebo Comparator)

INTERVENTIONS:
Behavioral: Physical activity counseling
  Arms: Exercise Counseling

SUMMARY:
This study aims at testing the efficacy of a physical activity (PA)intervention in an outpatient oncology setting. We plan to compare Brief Advice for PA (MD advice plus contact control) vs. Extended Advice (MD advice plus telephone-based PA counseling by research staff) over 3 months among 300 women who have completed treatment for breast cancer in the past 2 years.

Specific Aims: The primary aim is to examine the effects of oncologists' advice on PA plus telephone counseling (Extended Advice) vs. oncologists' advice (Brief Advice) alone on minutes of moderate-intensity PA at 3 months among 300 sedentary women who have completed treatment for breast cancer.

Secondary aims include examining a) the effects of the two interventions on participants' moderate-intensity PA at 6 and 12 months, b) the effects of the interventions on participants' physical functioning, fatigue, vigor and quality of life (QOL) at 3, 6 and 12 months, and c) the acceptability of the interventions to the oncologists and the usefulness of the interventions to patients.

DETAILED DESCRIPTION:
Background: With improved survival rates, there are growing numbers of cancer survivors. These individuals report impaired physical functioning, anxiety and depressed mood, fatigue, and reduced quality of life after treatment. In addition, they may be at increased risk for cardiovascular disease, obesity, osteoporosis and future cancers. Prior research has demonstrated that moderate-intensity physical activity (PA) can improve enhance physical functioning, reduce fatigue and improve vigor among cancer patients and those who have completed medical treatments. These efforts have not been integrated with the healthcare system. Data support the role of primary care providers in promoting PA among their sedentary patients; the role of oncologists in encouraging patients to become physically active has not been examined.

Objectives: This study aims at testing the efficacy of a PA intervention in an outpatient oncology setting. We plan to compare Brief Advice for PA (MD advice plus contact control) vs. Extended Advice (MD advice plus telephone-based PA counseling by research staff) over 3 months among 300 women who have completed treatment for breast cancer in the past 2 years.

Specific Aims: The primary aim is to examine the effects of oncologists' advice on PA plus telephone counseling (Extended Advice) vs. oncologists' advice (Brief Advice) alone on minutes of moderate-intensity PA at 3 months among 300 sedentary women who have completed treatment for breast cancer.

Secondary aims include examining a) the effects of the two interventions on participants' moderate-intensity PA at 6 and 12 months, b) the effects of the interventions on participants' physical functioning, fatigue, vigor and quality of life (QOL) at 3, 6 and 12 months, and c) the acceptability of the interventions to the oncologists and the usefulness of the interventions to patients.

Study Design: A randomized, controlled trial will be conducted in outpatient oncology practices in Rhode Island. Within this setting, the oncologists and research staff will offer a 3 month, theoretically-based intervention to increase moderate-intensity PA among 300 sedentary women aged 18 and older who attend cancer follow-up visits. The unit of randomization will be at the patient level.

Cancer Relevance: If the data are promising, the study lays the groundwork for improving cancer recovery by integrating a brief PA intervention into follow-up care for cancer survivors. This study offers the potential to improve the follow-up care for cancer survivors by encouraging them to becoming physically active, to help reduce the emotional and physical side-effects of cancer and its treatment, as well as possibly reduce their risk for other chronic diseases such as cardiovascular disease and osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

1) female aged >18 years, 2) completed primary and adjuvant treatment for breast cancer (patients on hormone treatment such as Tamoxifen will be eligible). Women on chemotherapy will become eligible 6 months after treatment completion, and will remain eligible up to 10 years posttreatment; 3) <10 years since treatment completion, 4) able to read and speak English, 5) provide consent for medical chart review to extract disease and treatment variables, 6) able to walk unassisted, are 7) sedentary defined as: currently not meeting ACSM/CDC criteria (Pate et al, 1995) for moderate-intensity activity (>30 mins. per day on >5 days per week) or vigorous-intensity activity (>20 mins. on >3 days per week), and 8) have access to a telephone. -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2004-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Minutes of moderate-intensity PA at 3 months among 300 sedentary women who have completed treatment for breast cancer. | 3 months

SECONDARY OUTCOMES:
Secondary aims include examining a) the effects of the two interventions on participants' moderate-intensity PA at 6 and 12 months, b) the effects of the interventions on participants' physical functioning, fatigue, vigor and quality of life (QOL) at | 6 and 12 months for physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Bernardine Pinto, Ph.D., Principal Investigator — The Miriam Hospital
Locations (1):
- Centers for Behavioral and Preventive Medicine, Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Pinto BM, Papandonatos GD, Goldstein MG. A randomized trial to promote physical activity among breast cancer patients. Health Psychol. 2013 Jun;32(6):616-26. doi: 10.1037/a0029886. PMID 23730723
- [Derived] Pinto BM, Dunsiger S, Waldemore M. Physical activity and psychosocial benefits among breast cancer patients. Psychooncology. 2013 Oct;22(10):2193-9. doi: 10.1002/pon.3272. Epub 2013 Mar 15. PMID 23494869